CLINICAL TRIAL: NCT03083327
Title: Prophylactic Early Parenteral Nutrition in Patients Undergoing Hematopoietic Cell Transplantation: A Multi-centre Randomised Controlled Trial.
Brief Title: Prophylactic Early PN in HPT/BMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sydney (Other)
Collaborators: Australasian Bone Marrow Transplant Recipient Registry (Unknown); University of Roma La Sapienza (Other); Northern Clinical School Intensive Care Research Unit, University of Sydney (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NHMRC APP1108301; ACTRN12615001329550 (Registry Identifier: Australian New Zealand Clinical Trials Registery); U1111-1194-5952 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2017-03-08; First posted 2017-03-20 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Parenteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessment of bone marrow biopsy to determine transplant success will be undertaken independent of the knowledge of treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): The control group in this study is pragmatic standard nutrition care. Currently after a bone marrow transplant in Australia, patients are normally fed orally for as long as possible. If oral intake fails to provide sufficient calories for a period of two to three days, enteral or parenteral nutrition may be provided.
  Interventions: Other: Pragmatic standard care.
- Early supplemental parenteral nutrition (Active Comparator): Supplemental prophylactic early parenteral nutrition will be commenced 1 day prior to conditioning chemoradiotherapy in patients who are not already malnourished. Supplemental parenteral nutrition continues throughout conditioning chemoradiotherapy and stem cell transplant.
  The dose of supplemental parenteral nutrition will be dependent on the total calories also received from oral and/or enteral nutrition intake.
  Interventions: Dietary Supplement: Parenteral nutrition.; Other: Pragmatic standard care.

INTERVENTIONS:
Dietary Supplement: Parenteral nutrition. — Nutrition support will be provides as per usual, but oral and enteral intake will be topped up with a standard parenteral nutrition solution. The standard parenteral nutrition solution will contain approximately 40 grams of amino acids/L, 40 g lipids/L and 100g dextrose/L).
  Arms: Early supplemental parenteral nutrition
Other: Pragmatic standard care. — Nutrition support will be provided as per usual care.

SUMMARY:
Supplemental prophylactic early parenteral nutrition will be commenced 1 day prior to conditioning chemoradiotherapy in patients who are not already malnourished. Supplemental parenteral nutrition continues throughout conditioning chemoradiotherapy and stem cell transplant.

DETAILED DESCRIPTION:
A standard parenteral nutrition solution will be used. The parenteral nutrition solution will be given once daily, and infused intravenously. The standard parenteral nutrition solution will contain approximately 40 grams of amino acids/L, 40 g lipids/L and 100g dextrose/L). Nutritional targets will be measured using indirect Calorimetry where available, or calculated via the Harris Benedict or Schofield equations. The dose of parenteral nutrition administered will be determined by the treating dietitian, treating physician or treating research team. The parenteral nutrition dose given will be individualised considering the patients clinical condition and body weight. The dose of supplemental parenteral nutrition will be dependent on the total calories also received from oral and/or enteral nutrition intake.

Supplemental parenteral nutrition will be discontinued when a patient is well enough to be discharged from hospital or when the patients attending clinician determines a central line is no longer needed for standard care. There is no maximum duration of supplemental parenteral nutrition..

Adherence to the study intervention will be monitored via medical chart reviews during site monitoring visits, and data queries on individual patient case report form documentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are about to commence conditioning chemoradiotherapy for allogeneic haematopoietic progenitor/stem cell transplantation, who have a haematological malignancy, who are not meeting 80% of their Caloric needs via oral or enteral intakes, and who are not malnourished.

Exclusion Criteria:

* Patients who are already receiving parenteral nutrition at time of screening.
* Patients with a documented licensing contraindication to parenteral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will be assigned a biological sex based on their legal gender established at time of enrolment.
Enrollment: 408 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival time | Recruitment will run for 3 years, with a median follow-up time of 2 years.
  Defined as time to relapse or death whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Gordon S Doig, PhD, Principal Investigator — Northern Clinical School Intensive Care Research Unit, University of Sydney
Locations (3):
- Australia (2):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Christchurch Hospital, CDHB, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided